CLINICAL TRIAL: NCT04273126
Title: Strengthening Homeless Families
Brief Title: Helping Families Pilot of a Family Resilience Program for Families Experiencing Homelessness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); American Academy of Child Adolescent Psychiatry. (Other)
Responsible Party: Principal Investigator, Roya Ijadi-Maghsoodi, MD, MSHPM, Assistant Professor in Residence, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: K12DA000357 (NIH); K12DA000357 (NIH)
Record Dates: First submitted 2020-01-22; First posted 2020-02-17 (Actual); Last update posted 2024-06-12 (Actual); Status verified 2024-06

CONDITIONS: Family Relationship; Coping Skills
Keywords: resilience, psychological; homelessness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): This arm consists of approximately 8-10 modules lasting approximately one hour and consisting of psychoeducation and core components including communication, problem solving, goal setting, and dealing with stress, tailored to families with experiences of homelessness and parental substance use.
  Interventions: Behavioral: Adapted Family Resilience Intervention

INTERVENTIONS:
Behavioral: Adapted Family Resilience Intervention — The program consists of approximately 8-10 modules lasting approximately one hour. Sessions focus on psychoeducation and key resilience skills.

SUMMARY:
The goal of this study is to pilot an adapted family resilience program among families with a recent history of homelessness in Los Angeles County and to assess for feasibility and acceptability. The investigators have adapted a family resilience program called Families Overcoming Under Stress (FOCUS), a trauma-informed intervention designed for families experiencing trauma, parental substance use, and homelessness. Our primary hypothesis is that the adapted family resilience program will be feasible and acceptable to families with a recent history of homelessness. Families that are eligible to participate in the study will be assigned to the adapted family resilience intervention. The intervention program consists of around 8-10 modules lasting up to one hour each. The program provides psychoeducation and teaches resilience skills including communication, problem solving, goal setting, and how to deal with stress. Families will be asked to fill out 3 surveys (one at the beginning of the program, one at the end of the program, and at 6 months follow-up). Some families may also be asked to participate in a hour long interview after the completion of the program for feedback on the program.

At this time, all assessments and intervention are being conducted remotely due to the pandemic.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Family has a history of homelessness within the past two years (homelessness defined by the Department of Health and Human Services definition)
* Parent/guardian/caregiver has custody of and cares for a youth between the ages of 8-17
* Both youth and parent/guardian/caregiver are able to take part in an 8 module session intervention

Exclusion Criteria:

* Does not meet inclusion criteria
* Has taken part in a Families OverComing Under Stress (FOCUS) intervention previously

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2020-02-19 (Actual); Primary Completion 2023-04-03 (Actual); Study Completion 2023-04-03 (Actual)

PRIMARY OUTCOMES:
Feasibility of the adapted family resilience intervention for families experiencing homelessness and parental SUDs through retention rates of participants. | 6 months
  Feasibility is defined as the extent to which the adapted intervention can be implemented with families with an experience of homelessness and parental SUDs, assessed through measuring rate of retention of participants.
Feasibility of the adapted family resilience intervention for families experiencing homelessness and parental SUDs through completion of program core components. | 3 months
  Feasibility is defined as the extent to which the adapted intervention can be implemented with families with an experience of homelessness and parental SUDs, assessed through measuring number of program core components completed by participants.
Acceptability of the adapted family resilience intervention to families experiencing homelessness and parental SUDs through qualitative interviews with youth and parents inquiring about intervention acceptability. | 3 months
  The investigators will assess acceptability of implementing the adapted intervention with families experiencing homelessness and parental SUDs by conducting qualitative interviews with a subset of parent and youth participants completing the intervention. The interviews will explore acceptability of the intervention to families experiencing homelessness and parental substance use disorders and recommendations for improvement. The interviews will be audio-recorded, transcribed, and analyzed using thematic content analysis.
Acceptability of the adapted family resilience intervention through a self-report intervention acceptability measure. | 3 months
  Acceptability is defined as the perception that the adapted intervention is agreeable and satisfactory.The investigators will administer a self-report measure of the acceptability of core components of the intervention to be completed following the intervention by parents and youth, with higher score indicating greater acceptability of the intervention to families experiencing homelessness and parental SUDs. Each individual item is scaled with a range of 1 (low) to 5 (high).

SECONDARY OUTCOMES:
Alcohol, Smoking, and Substance Involvement Screening Test (ASSIST) | Baseline, 3 month, 6 month
  Self reported measure administered to parents in the study to assess for substance use across lifetime and in the past 3 months. Each of the 8 item responses vary in scoring. The total substance involvement score (global continuum of risk) can be calculated by summing up the responses to all items. A higher score indicates higher risk for problems related to substance use.
Addiction Severity Index (ASI) | Baseline, 3 month, 6 month
  Self reported measure administered to parents to assess for drug and alcohol use in the past 30 days and lifetime of regular use. The ASI does not yield a composite score but assesses days of use and extended periods of use.
General Anxiety Disorder (GAD-7) | Baseline, 3 month, 6 month
  Self reported measure administered to parents to assess anxiety level. Each of the 7 item responses are scored from 0 (not at all) to 3 (nearly every day), yielding a total score ranging from 0-21. A higher score suggests higher level of anxiety.
Patient Health Questionnaire (PHQ-9) | Baseline, 3 month, 6 month
  Self reported measure administered to parents to assess depression severity. Each of the 9 item responses are scored from 0 (not at all) to 3 (nearly every day), yielding a total score ranging from 0-27. A higher score suggests higher level of depression.
PTSD Checklist for the DSM-V (Diagnostic and Statistical Manual) | Baseline, 3 month, 6 month
  Self-reported measure administered to parents that assesses the severity of PTSD symptoms over the past month. The PTSD Checklist for DSM-5 (PCL-5), the responses are scored from 0 (not at all) to 4 (extremely). To assess total symptom severity, scores for each of the 20 items are summed, the range is 0-80, with higher levels indicating higher severity.
Short Form 12 (SF-12) | Baseline, 3 month, 6 month
  Self reported measure administered to parents to assess health and well-being. The SF-12 is scored as physical (PCS-12) and mental (MCS-12) component summary scales. The PCS-12 and MCS-12 scores use norm-based scoring with 50 being the population mean. The possible scores for PCS-12 and MCS-12 could range from 0 (worst) to 100 (best), with scores above and below 50 being above and below average.
Connor-Davidson Resilience Scale (CD-RISC) | Baseline, 3 month, 6 month
  Self reported measure administered to parents to assess resilience. Each of the 10 item responses are scored from 0 (not true at all) to 4 (true nearly all of the time), yielding a total score that ranges from 0-40. A higher score indicates more resilience.
Medical Outcomes Study Social Support Survey (MOS-SSS) | Baseline, 3 month, 6 month
  Self-reported measure administered to parents to assess social support. Each of the of 8 item responses are scored from 1 (none of the time) to 5 (all of the time), yielding a total score that ranges from 8-40. A higher score for an individual scale or for the overall support index indicates more support.
Monitoring the Future Scale (Substance Use Scale) | Baseline, 3 month, 6 month
  Self reported measures to assess substance use in the past 30 days and lifetime for youth for each selected substance. For the 29 items, responses range from from "0 occasions of use" to "40 or more occasions of use."
Monitoring the Future Scale (Perceived Risk Scale) | Baseline, 3 month, 6 month
  Self reported measure to assess perceived risks of substance use for youth for each selected substance. For the 6 items, each response ranges from "no risk" to "great risk", with the option to select "can't say, drug unfamiliar."
Monitoring the Future Scale (Disapproval Scale) | Baseline, 3 month, 6 month
  Self reported measure to assess disapproval of substance use for youth. For each of the 17 items, responses range from "not disapprove" to "strongly disapprove."
Strength and Difficulties Questionnaire (SDQ) | Baseline, 3 month, 6 month
  Self reported measure to assess psychological strengths and difficulties of children/youth. Parents will complete the measure for their children. The measure will also be delivered to youth (age 11-14). Each of the 25 item responses are scored from 0 (not true) to 2 (certainly true). The items are divided into 5 subscales (emotional problems, conduct problems, hyperactivity, peer problems, and prosocial). The first four subscales refer to difficulties that children may have and may be group together in a general subscale of difficulties (20 items). The subscale of prosocial skills refer to positive and adaptive behaviors. For each of the 5 subscales, the score can range from 0-10. The score of the difficulties subscale ranges from 0 to 40. Higher scores suggest higher emotional and behavioral symptoms.
Screen for Child Anxiety Related Emotional Disorders (SCARED) | Baseline, 3 month, 6 month
  Self reported measure to assess childhood anxiety disorders, including panic, generalized anxiety, separation anxiety, social phobia, and school phobia among children . Each of the 41 item responses are scored from 0 (not true or hardly ever true) to 2 (very true or often true), yielding a total score ranging from 0-82.
Mood and Feelings Questionnaire (MFQ) | Baseline, 3 month, 6 month
  Self reported measure to assess depression in children and youth. Each of the 13 item responses are scored from 0 (not true) to 2 (true), yielding a total score ranging from 0-26. A higher score suggests more severe depressive symptoms.
Resistance to Peer Influence Scale | Baseline, 3 month, 6 month
  Self reported measure to assess resistance to peer influence for youth.The measure presents respondents with a series of 10 pairs of statements and asks them to choose the statement that is the best descriptor. After indicating the best descriptor, the respondent is then asked whether the description is "Really True" or "Sort of True." Responses are then coded on a 4-point scale, ranging from "Really true" for one descriptor to "Really true" for the other descriptor, and averaged. A higher score suggests greater resistance to peer influence.
Children's Coping Strategies Checklist-Revision 1 (CCSC-R1) | Baseline, 3 month, 6 month
  Self reported measure to assess coping strategies among youth. Each of the 54 item responses are scored from 1 (never) to 4 (always). Scoring for the four major factors of coping is reached by taking the mean.
Resilience Youth Development Module (RYDM) of the California Healthy Kids Survey (CHKS) | Baseline, 3 month, 6 month
  Self reported measure to assess internal assets for children and youth. Each of the 12 item responses are scored from 1 (not at all true) to 4 (very much true), yielding a score that ranges from 12 to 48. A higher score indicates higher levels of internal assets.
Deviant Peer Affiliation Scale | Baseline, 3 month, 6 month
  Self reported measure to assess deviant peer affiliations for youth (age 12-14). Each of the 3 item responses are scored from 1 (very few) to 5 (almost all), with the exception of one reverse-coded item. The total score is computed by averaging across all items. A higher score suggests greater deviant peer affiliations.
McMaster Family Assessment Device (FAD) | Baseline, 3 month, 6 month
  Self reported measure to assess family functioning for parents and youth over 12. Each of the 12 item responses are scored from 1 (strongly agree) to 4 (strongly disagree). The scores are added up and then divided by the number of items, giving a total score ranging from 1 to 4. A higher score indicates worse functioning.
Parental Sense of Competence Scale (PSOC) | Baseline, 3 month, 6 month
  Self reported measure for parents to assess parenting self-esteem. Each of the 17 item responses are scored from 1 (strongly disagree) to 6 (strongly agree), yielding a total score that ranges from 17-102. A higher score suggests greater self-esteem.
Parental Monitoring Scale | Baseline, 3 month, 6 month
  Self reported measure to assess adolescents' perception of their parents' monitoring. Each of the 6 item responses are scored from 1 (never) to 5 (always). A composite score is obtained by averaging responses to the 6 items. A higher score indicates higher perceived perception of parent monitoring. This scale is also delivered to parents, in order to assess the parent's perception of their supervision. A composite scale score is obtained in the same manner. Higher score indicates higher perceived perception of their monitoring.

CONTACTS AND LOCATIONS:
Overall Officials: Roya Ijadi-Maghsoodi, MD, MSHPM, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No